CLINICAL TRIAL: NCT02840357
Title: The Purple Wheat Intervention Study: Impact of Purple Wheat Consumption on Markers of Inflammation and Oxidative Stress in Adults.
Brief Title: Impact of Purple Wheat Consumption on Markers of Inflammation and Oxidative Stress in Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Amanda Wright, Ph.D, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PWIS2
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Chronic inflammation; Adults; overweight; obese
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): Purple Wheat Convenience Bars The treatment group will consume 4 servings /day of bran-enriched purple wheat convenience bars (40g/ serving)
  Interventions: Other: Purple Wheat Convenience Bars
- Control Group (Placebo Comparator): Control Wheat Convenience Bars The control group will consume 4 servings /day of bran-enriched ordinary wheat convenience basr (40g/ serving)
  Interventions: Other: Control Wheat Convenience Bars

INTERVENTIONS:
Other: Purple Wheat Convenience Bars — Whole grain convenience bars manufactured with purple wheat
  Arms: Treatment Group
Other: Control Wheat Convenience Bars — Whole grain convenience bars manufactured with ordinary wheat
  Arms: Control Group

SUMMARY:
The main purpose of this study is to determine the effect of consumption of purple wheat anthocyanin-rich products for eight weeks by human participants with an elevated level of chronic inflammation, on oxidative stress and inflammatory responses as measured by select plasma biomarkers.

DETAILED DESCRIPTION:
This study will investigate the effect of daily consumption of purple wheat bran-enriched wholegrain convenience bars, for 8 weeks on inflammation and oxidative stress biomarkers and plasma antioxidant capacity. This study is a randomized, parallel arm study with 20 men and 20 women who will adhere to a low anthocyanin and low phenolic aid diet for the duration of the study. The participants will be randomly divided into two groups, using stratification for matching sex and screening hs-CRP level to be equally distributed in each group, and assigned to either the treatment group or control group. Both group will have a 10 day diet run-in period where consumption of foods rich in anthocyanins and phenolic acids will be limited. Both groups will consume 4 servings of wheat products per day for 8 weeks and will replace 4 grain servings from their typical daily intake with the study treatment products. Fasting blood samples will be collected during three study visits, including baseline, for the analysis of inflammatory and oxidative stress biomarkers and plasma antioxidant capacity. The plasma metabolites of anthocyanins and phenolic acids will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2 and/or Waist circumference ≥102 cm (men) and ≥88 cm (women)
* hs-CRP: ≥ 1.0 mg/L at time of screening
* Stable (>3 months) and consistent use of all prescribed medications and/or supplements
* Non- to moderate alcohol consumer (i.e. less than 5 drinks per sitting and no more than 14 per week)
* Not taking any antibiotics within the last 3 months, or planning to take antibiotics within the next 6 months

Exclusion Criteria:

* Pregnant or breastfeeding females
* Lifetime history of any acute medical event, including but not limited to, heart attack or stroke
* Occasional or intermittent smoker (includes but not limited to tobacco and cannabis)
* Consistent smoker of <1 year
* Recent diagnosis (within 6 months) of a serious medical condition, including but not limited to, cancer, diabetes, heart disease or hepatitis
* Recent history (within 6 months) of a clinically significant psychiatric disorder, other than mild depression
* Any disorder of the gastrointestinal system or food intolerances, including but not limited to, inflammatory bowel disease or Celiac disease
* Any food allergies or any life-threatening allergies, food or otherwise
* Regular recreational drug use of more than once per week, including but not limited to cannabis, magic mushrooms, ecstasy etc
* Difficulty providing blood samples

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Serum concentration of inflammatory biomarker (hs-CRP) | Fasting (0 hours)

SECONDARY OUTCOMES:
Plasma concentration of lipids | Fasting (0 hours)
Plasma concentration of inflammatory biomarkers | Fasting (0 hours)
Plasma concentration of total antioxidant capacity | Fasting (0 hours)
Plasma concentrations of anthocyanin metabolites and phenolic acids | Fasting (0 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, University of Guelph, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Through peer reviewed publications.